CLINICAL TRIAL: NCT02526004
Title: Cystic Fibrosis Microbiome-determined Antibiotic Therapy Trial in Exacerbations: Results Stratified
Acronym: CFMATTERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Queen's University, Belfast (Other); University of Paris 5 - Rene Descartes (Other); University of Dundee (Other); University of Washington (Other); University Hospital Heidelberg (Other); Teagasc (Industry); Clininfo S.A. (Industry); GABO:mi (Industry); Papworth Hospital NHS Foundation Trust (Other Government); KU Leuven (Other); Assistance Publique - Hôpitaux de Paris (Other); European Union (Other)
Responsible Party: Principal Investigator, Barry Plant, Barry Plant, CFMATTERS Coordinator, University College Cork
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: UCC-CFMATTERS
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Microbiome; Stratified Antibacterial therapy; Resistance; Pathogen Host Interaction
MeSH Terms: conditions — Cystic Fibrosis | interventions — Ceftazidime; Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Empiric Treatment (Active Comparator): Ceftazidime or Aztreonam (in case of Ceftazidime allergy) and Tobramycin
  Interventions: Drug: Ceftazidime; Drug: Tobramycin
- Microbiome Guided Treatment (Experimental): Ceftazidime or Aztreonam (in case of Ceftazidime allergy) and Tobramycin and 3rd Antibiotic based on the Microbiome analysis
  Interventions: Drug: Ceftazidime; Drug: Tobramycin

INTERVENTIONS:
Drug: Ceftazidime
Drug: Tobramycin

SUMMARY:
Antimicrobial resistance is a significant challenge facing global healthcare. The unnecessary use of antibiotics is a key driver in the development of antibiotic resistance. Cystic Fibrosis (CF) represents a unique disease model to study bacterial resistance and to explore therapeutic strategies for same, as chronic lung infection overlaps with acute lung exacerbation's caused by a multitude of organisms. With time, chronic polymicrobial infection develops, with the most dominant infecting organism being Pseudomonas aeruginosa. In acute CF infections, empiric intravenous antibiotics are usually given for two weeks. Recurrent infections and treatments result in increasing antimicrobial resistance, and alterations in pathogen host interactions in the lung and gut flora. Next-generation DNA sequencing technology now offers DNA-based personalised diagnostics and treatment strategies. Enhancing our knowledge of the microbiome allows the use of stratified targeted antibacterial therapy that can be compared with standard empirical antibacterial therapy currently used. Cystic Fibrosis Microbiome-determined Antimicrobial Therapy Trial in Exacerbations: Results Stratified (CFMATTERS) will provide a randomized multi-centre controlled trial of microbiome-derived antimicrobial treatments versus current empirical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written and informed consent, and assent where required.
* Age 16 years or older at enrolment
* Diagnosis of CF by standard sweat test and/or genetic analysis
* Persistent pulmonary Pseudomonas aeruginosa colonization confirmed on at least 2 occasions in the preceding 12 months
* Screening FEV1 predicted of >25%
* Able to perform spirometry reproducibly prior to enrolment
* Able to expectorate and provide a sputum sample at least once daily
* ≥1 non-elective course of intravenous antibiotics in the preceding year
* Able to understand and comply with protocol requirements, restrictions and instructions and likely to complete the study as planned, as judged by the investigator

Exclusion Criteria:

* Life expectancy less than 6 months
* They are a solid organ transplant recipient
* Have a requirement for immunosuppression ≥10mg corticosteroids per day
* Previous positive culture of non-tuberculosis mycobacteria species M.avium, M.abscessus or M.intracellulare within the last 12 months or undergoing active therapy
* Positive culture of any Burkholderia cepacia species within the last 12 months or undergoing active therapy
* Allergic bronchopulmonary aspergillosis on treatment
* Known allergies to more than 3 different classes of antibiotics, and intolerance or allergy to tobramycin.
* Liver portal hypertension, determined by identification of oesophageal varices
* Advanced kidney disease requiring a dose reduction of ceftazidime or contraindicating aminoglycosides
* History of any illness that in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject
* If patient undergoes a pulmonary exacerbation before the Microbiome analysis is reviewed by the Consensus Treatment Panel and i.v. antibiotics are administered. In this case, a repeat sputum will be sent for analysis 4 weeks after end of antibiotic treatment.
* Pregnant or breast-feeding at time of eligible pulmonary exacerbation

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
The percentage change in recovery (post-exacerbation) FEV1 relative to the previous pre-exacerbation FEV1. | Time from enrollment to 14 days post initiation of IV antibiotics for elligible exacerbation.

SECONDARY OUTCOMES:
The time to next pulmonary exacerbation | Time from pulmonary exacerbation day 0, to next pulmonary exacerbation up to study close month 21
The improvement in symptom burden by day 7 as determined by Cystic Fibrosis Respiratory Symptom Diary (CFRSD) | Time from pulmonary exacerbation day 0 to day 7 of pulmonary exacerbation
  As determined by Cystic Fibrosis Respiratory Symptom Diary (CFRSD)
The improvement in health related quality of life at day 28 post treatment and at 3 months as determined by the Cystic Fibrosis Questionnaire Revised (CFQR) | Time from pulmonary exacerbation day 0 to day 28 and month 3 post study treatment
  As determined by the Cystic Fibrosis Questionnaire Revised (CFQR)
Total number of i.v. antibiotic days (home or in hospital) from time of randomisation in the trial | Time from enrollment in the study up to study close month 21
Change in FEV1 | Time from enrollment in the study up to study close month 21
Total number of exacerbations post trial treatment | Time from pulmonary exacerbation day 0 to study close month 21

CONTACTS AND LOCATIONS:
Locations (1):
- University College Cork, Cork, Cork, Ireland